CLINICAL TRIAL: NCT02254811
Title: A Prospective, Multi-center, Randomized Trial of Fecal Microbiota Transplantation (FMT) Delivered by Capsule vs Colonoscopy in the Management of Recurrent Clostridium Difficile Infection (CDI)
Brief Title: FMT Delivered by Capsule Versus Colonoscopy for Recurrent C. Diff
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Dina Kao, Associate Professor, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48233
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Enterocolitis Clostridium Difficile Recurrent
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delivery via capsule (Experimental): Fecal microbiota transplant is delivered by oral capsules
  Interventions: Biological: Fecal Microbiota Transplant
- Delivery via colonoscopy (Experimental): Fecal microbiota transplant delivered by colonoscopy
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — transfer of healthy human gut bacteria to restore the microbiome

SUMMARY:
Delivery of FMT by upper route, including gastroscopy, nasogastric/ nasojejunal tube, and lower route, including retention enema, sigmoidoscopy, or colonoscopy have all been utilized successfully. Endoscopic delivery requires significant health care utilization and associated cost. Therefore, it is extremely desirable if FMT can be infused by a non invasive modality, which would significantly reduce patient discomfort, procedure related risks and health care costs, while offering similar efficacy to colonoscopic delivery in the range of 90%.

DETAILED DESCRIPTION:
Patients with minimum 3 episodes of Clostridium difficile within 6 months are randomized 1:1 to received FMT by either colonoscopy or capsules. Pts are assessed at 1 week, 2 weeks, 1 mon, 3 mon, 6 mon and 1 year post FMT. Stool, urine and blood samples are collected. Medical cost for previous treatment is collected as well at pt perspective and QoL.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 90 years at the time of Screening.
2. Diagnosis of at least 3 episodes of recurrent CDI, with each episode defined as presence of diarrhea (> 3 unformed stools/24 hours) associate with positive stool Clostridium difficle toxin, occurring within 3 months of each other.
3. CDI infection under symptomatic control with < 3 loose/unformed BM's per 24 h period for at least 2 consecutive days before procedure.
4. Those with ability to provide informed consent.

Exclusion Criteria:

1. Those with complicated CDI, defined as white blood cell>35 or <0.5 x 109/L, significant abdominal pain and distension with evidence of toxic megacolon or pseudomembranous colitis, hypotension defined as systolic blood pressure < 90 mmHg unresponsive to fluid resuscitation, end organ failure, or requiring intensive care unit admission.
2. Those with chronic diarrheal illness, such as irritable bowel syndrome or inflammatory bowel disease unless they are in remission for at least 3 months prior to enrollment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients without recurrent CDI | 12 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dina Kao, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kao D, Roach B, Silva M, Beck P, Rioux K, Kaplan GG, Chang HJ, Coward S, Goodman KJ, Xu H, Madsen K, Mason A, Wong GK, Jovel J, Patterson J, Louie T. Effect of Oral Capsule- vs Colonoscopy-Delivered Fecal Microbiota Transplantation on Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2017 Nov 28;318(20):1985-1993. doi: 10.1001/jama.2017.17077. PMID 29183074